CLINICAL TRIAL: NCT02809131
Title: Randomized Noninferiority Study of an Antibacterial Envelope Alone Versus Envelope Plus Intraoperative Antibacterial Irrigant and Postoperative Antibiotics to Prevent Cardiac Implantable Electronic Device Infections in High-Risk Patients
Brief Title: Perioperative Antibiotic Therapy to Prevent Cardiac Implantable Electronic Device Infections.
Acronym: ENVELOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Thomas Jefferson University (Other); The Cooper Health System (Other); Valley Health System (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Christopher Ellis, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150753
Record Dates: First submitted 2016-04-27; First posted 2016-06-22 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Sick Sinus Syndrome; Complete Heart Block; Syncope; Chronic Systolic Heart Failure
Keywords: CIED infection
MeSH Terms: conditions — Sick Sinus Syndrome; Syncope | interventions — Bacitracin; Cephalexin; Levofloxacin; Clindamycin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline irrigation (Experimental): Saline irrigation
  Interventions: Drug: Saline
- Antibiotic irrigation and PO antibiotics (Active Comparator): Antibacterial irrigant (polymyxinB/bacitracin) and postoperative oral antibiotics (cephalexin, clindamycin, or levofloxacin)
  Interventions: Drug: polymixin/bacitracin; Drug: cephalexin, or levofloxacin, or clindamycin

INTERVENTIONS:
Drug: polymixin/bacitracin — Antibacterial irrigation
  Arms: Antibiotic irrigation and PO antibiotics
Drug: cephalexin, or levofloxacin, or clindamycin — Post operative oral antibiotics
  Other Names: Kelfex, Levaquin, Cleocin
  Arms: Antibiotic irrigation and PO antibiotics
Drug: Saline — Saline irrigation
  Arms: Saline irrigation

SUMMARY:
The number of cardiac implantable electronic devices (CIEDs) implanted each year has grown rapidly over the past two decades. CIED infections, defined as infections involving the generator implant site (pocket) and/or intravascular leads, have become increasingly prevalent, with the rate of growth in infections outpacing that of CIED procedures. The odds of both short term and long term mortality are at least doubled in patients who suffer CIED infections, and long term survival is particularly poor in women. Optimal strategies to prevent CIED infections in high-risk patients are largely unproven. However, recent observational studies of an antibiotic-coated envelope implanted at the time of CIED procedure have shown that this strategy is associated with a low incidence of CIED infections. Other interventions to prevent CIED infections, including the use of antibiotic irrigant used to wash the pocket during implantation and postoperative oral antibiotics, are commonly used but not supported by rigorous controlled studies. The Specific Aim of this study is to test the hypothesis that the use of the antibacterial envelope alone is noninferior to a strategy using the antibacterial envelope and intraoperative antibacterial irrigant and postoperative oral antibiotics for the reduction of cardiac implantable device infections in patients with ≥2 risk factors for infection.

DETAILED DESCRIPTION:
1.0 Background

The number of cardiac implantable electronic devices (CIEDs) implanted each year has grown rapidly over the past two decades, largely due to expanding use of implantable cardioverter-defibrillators (ICDs) and devices capable of delivering cardiac resynchronization therapy (CRT). CIEDs have increasingly been utilized in older patients with multiple medical comorbidities. As a result CIED infections, defined as infections involving the generator implant site (pocket) and/or intravascular leads, have become increasingly prevalent, with the rate of growth in infections outpacing that of CIED procedures. The increase in incidence of CIED infections has outpaced the growth in device implantation, in large part due to the medical complexity of today's CIED patients. These devastating complications are associated with significant cost, morbidity, and mortality. The odds of both short term and long term mortality are at least doubled in patients who suffer CIED infections, and long term survival is particularly poor in women.

Patient-specific risk factors for CIED infections have been examined in multiple registries and case-control studies. For patients with at least two risk factors, the reported incidence of CIED infection is 2-3%. Management of these infections is complex and expensive. The cornerstone of management is the complete removal of all infected hardware whenever possible, which in itself poses significant risks for patients. Therefore prevention of infections is crucial.

Best practices for reducing CIED infections are an active area of research. Since most infections occur as a result of bacterial seeding at the time of device implantation or revision, careful attention to strict sterile technique is mandatory. Optimal skin preparation and perioperative intravenous antibiotics have been associated with a reduced rate of CIED infections in randomized controlled studies. Additionally, several recent retrospective studies have suggested an important role of the minocycline and rifampin impregnated TYRX antibacterial envelope in reducing infections. The device consists of 2 polypropylene mesh sheets joined on 3 sides with a 3mm seam and is available in 2 sizes to accommodate pacemaker and ICD pulse generators. This polypropylene envelope releases minocycline and rifampin from a bioresorbable polyarylate polymer over approximately 7 days, directly into the CIED generator pocket.

Aside from optimal skin preparation and perioperative intravenous antibiotics, other practices to reduce the risk of CIED infections vary widely. Many operators use an antibacterial solution (e.g., polymyxin-B/bacitracin) to irrigate the pocket during device implantation. Additionally, many centers have adopted the routine use of prophylactic postoperative antibiotics to reduce the risk of CIED infections. However, neither of these strategies has been evaluated in randomized clinical studies. Antibacterial irrigation solution is expensive, and oral antibiotics are associated with a small yet clinically important risk of adverse effects, including Clostridium difficile infection. Therefore, prospective randomized studies are needed to evaluate the efficacy, safety, and cost-effectiveness of intraoperative antibacterial rinse and postoperative oral antibiotics.

Summary of significance: CIED infections constitute major complications of device implantations or revisions and are becoming increasingly prevalent. Infections are associated with increased morbidity, mortality, and cost, and are very difficult to treat. Recent studies have explored ways to reduce the incidence of CIED infections, and use of the TYRX antibacterial envelope has emerged as a potential strategy for prevention. Other strategies including intraoperative antibacterial irrigation and postoperative oral antibiotics are commonly used despite the lack of prospective studies documenting efficacy, safety, and cost-effectiveness. We and others have reported a very low incidence (<1%) of CIED infections in high-risk patients receiving the TYRX antibacterial envelope. One intriguing possibility is that the antibacterial envelope can be used instead of intraoperative antibacterial rinse and postoperative oral antibiotics. Therefore, an important knowledge gap exists about the best practices to prevent CIED infections in high-risk individuals.

2.0 Rationale and Specific Aims

SPECIFIC AIM: to test the hypothesis that the use of the TYRX antibacterial envelope alone is noninferior to a strategy using the antibacterial envelope and intraoperative antibacterial irrigant and postoperative oral antibiotics for the reduction of cardiac implantable device infections in patients with ≥2 risk factors for infection.

CIED infections are devastating yet potentially preventable complications. We previously conducted a retrospective study of the TYRX antibacterial envelope and found that use of the device in patients with ≥2 risk factors for CIED infection was associated with a markedly decreased infection rate (0.4% with the device versus 3% without, adjusted odds ratio [95% confidence interval]: 0.09 [0.01 to 0.73], P =0.02). All patients in our previous study had intraoperative irrigation of the device pocket with polymyxin-B/bacitracin solution and received routine postoperative oral antibiotics consistent with local practices. However, whether use of intraoperative irrigant and postoperative antibiotics reduces the risk of infection has not been evaluated in prospective, randomized trials. Moreover, it is unknown whether these treatments offer any incremental benefit over the use of the TYRX antibacterial envelope alone.

Given the significant cost of polymyxin-B/bacitracin solution and concerns over unnecessary use of oral antibiotics and emerging resistant microorganisms, it is critically important to establish whether these treatments offer any incremental benefit for patients at high risk for a CIED infection who are receiving the TYRX antibacterial envelope. The Specific Aim of this study will be to prospectively test the hypothesis that an infection risk-reduction strategy using the TYRX antibacterial envelope alone is noninferior to a strategy using the envelope with intraoperative antibacterial irrigant and postoperative oral antibiotics in patients undergoing a CIED procedure who have at least 2 CIED infection risk factors.

3.0 Previous Animal and Human Studies

The TYRX antibacterial envelope effectively prevented CIED infections in an animal model. In an animal model of direct bacterial inoculation into the device pocket, the TYRX antibacterial envelope showed excellent activity against Staphylococcus epidermidis, Staphylococcus capitis, Escherichia coli, and Acinetobacter baumannii. Importantly, systemic levels of minocycline and rifampin were undetectable.

Use of the TYRX antibacterial envelope has been associated with a reduced incidence of CIED infections in retrospective studies of high-risk patients. In a multi-center trial, use of the TYRX antibacterial envelope was associated with a low risk of CIED infections (0.5%). However, the relatively short follow-up period (mean: 1.9 months) and lack of a control arm limited the interpretation of the study's results. We conducted a retrospective controlled study of the TYRX antibacterial envelope in patients with at least 2 CIED infection risk factors at our institution. Among 260 TYRX envelope recipients, the incidence of CIED infection after a mean 18.7 month follow-up period was 0.4%, compared with 3% in 639 high-risk controls who did not receive the envelope (adjusted odds ratio: 0.09, 95% confidence interval 0.01 to 0.73, P =0.02). Another retrospective study at a high-volume center found that the prevalence of CIED infections decreased from 1.5% to 0.6% after the TYRX antibacterial envelope was instituted into practice (P =0.03).

Based on these and other studies, the Worldwide Randomized Antibiotic Envelope CIED Infection Prevention Trial (WRAP-IT) was conceived. This landmark trial will prospectively evaluate the efficacy of the TYRX-A antibacterial envelope. However, our proposed study will be complementary to the WRAP-IT trial because we will specifically evaluate whether the TYRX-A antibacterial envelope alone offers ample protection against CIED infections without the use of intraoperative antibacterial solution and postoperative oral antibiotics.

6.0 Study Procedures

Device implantation and follow-up. CIED procedures will be performed in accordance with established practice guidelines. Perioperative procedures to reduce the risk of CIED infection including optimal skin preparation and intravenous antibiotics (cefazolin or vancomycin) will be applied to all patients. All patients will receive the TYRX absorbable antibacterial envelope. Patients randomized to the intraoperative antibacterial irrigant/postoperative oral antibiotic (control) arm will undergo irrigation of the device pocket with up to 1 liter polymyxin-B/bacitracin solution. Patients in the control arm will also receive 3 days of postoperative oral antibiotics (cephalexin 500mg 3 times daily, clindamycin 300mg 3 times daily, or levofloxacin 500mg once daily) as per investigator routine ordering practice with discretion per each individual patient. Patients randomized to the experimental arm will not receive intraoperative antibacterial irrigation (will be allowed up to 1 liter sterile saline irrigation), nor post-operative oral antibiotics.

All patients will be followed after their procedures according to established practice guidelines. At a minimum, patients will be seen 4 weeks after the procedure for a wound check, at 6 months, and then every year or more frequently as dictated by each patient's clinical status. A digital photograph of the device pocket will be captured at the 4-week postoperative visit. In addition, the study nurse will telephone each patient 3 months after implantation to assess for symptoms and signs of infection. For the purposes of the study, patients will continue to be followed for a minimum of 6 months after the procedure, but additional follow-up data after six months may be collected continuously until the study closes.

Ascertainment of the primary endpoint: CIED infection after a minimum 6-month follow-up period. The primary study endpoint will be CIED infection resulting in complete CIED system removal, antibiotic therapy in patients who are not candidates for system removal, or death due to CIED infection. To avoid detection bias we will prospectively apply criteria for definition of the primary endpoint and ask treating physicians to thoroughly document objective findings.

Examples of objective signs of CIED infection.

Objective findings of CIED infection

* Fever or leukocytosis without an alternative explanation (e.g., urinary tract infection or pneumonia)
* Tenderness, erythema, or warmth at the pulse generator site
* Purulent discharge from the pulse generator site (from incision or fistula)
* Positive blood or pulse generator site cultures
* Vegetation adherent to CIED hardware
* Purulent material within pulse generator pocket upon reoperation

A digital photograph of the device pocket will be captured routinely at the postoperative visit and whenever CIED infection is a consideration. In case of a suspected CIED infection, treating physicians will be strongly encouraged to obtain peripheral blood cultures prior to initiation of antibiotic therapy and intraoperative cultures during CIED system removal. A panel of 3 physicians at the coordinating center who are blinded to study assignment (experimental versus control) will independently adjudicate outcomes in "real time" and will vote whether or not the criteria for CIED infection have been met. A minor superficial infection of the incision that does not involve the generator pocket, does not result in any systemic symptoms or signs, and is treated with either observation or a short course of oral antibiotics, will not be counted as a CIED infection but will be considered a secondary endpoint.

Study oversight: The principal investigator at each study sight will be responsible for all aspects of the study at their respective sites. To ensure fidelity with the study protocol, an independent study coordinator at Vanderbilt University who is not directly involved with the study will review upon initiation of the study and first patient enrolled at each site, and then a random selection (10%) of patient records at each site (including Vanderbilt University) on a continuous basis set out by the monitoring agreement throughout the duration of the study, and quarterly prepare a report for the study's principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Able to give informed consent
* At least 2 of the following risk factors for infection:

  * Diabetes mellitus
  * Chronic kidney disease (estimated creatinine clearance <30 ml/min
  * Therapeutic anticoagulation
  * Chronic heart failure
  * Chronic use of corticosteroids
  * Fever ≥38° C or leukocytois (≥11,000 cells/mm3) within 24 hrs of implant
  * Device revision (including generator change, or extraction)
  * ≥3 leads in situ (CRT system or abandoned leads)
  * Early reoperation (pocket re-entry <2 weeks)
  * Previous CIED infection

Exclusion Criteria:

* Medical condition that is likely to be fatal in less than one year
* Emergent CIED procedure
* Allergy to rifampin or minocycline, Allergy to polymyxin-B or bacitracin
* Enrollment in WRAP-IT trial
* Current CIED pocket infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ellis, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellis CR, Greenspon AJ, Andriulli JA, Gould PA, Carillo RG, Kolek MJ, Donegan R, Amaral AP, Mittal S. Randomized Trial of Stand-Alone Use of the Antimicrobial Envelope in High-Risk Cardiac Device Patients. Circ Arrhythm Electrophysiol. 2023 May;16(5):e011740. doi: 10.1161/CIRCEP.122.011740. Epub 2023 Mar 24. PMID 36960716

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Irrigation: Saline Irrigation in patients undergoing a cardiac implantable electronic devices (CIED) procedure who have at least 2 CIED infection risk factors
- Antibiotic Irrigation and Oral Antibiotics: Antibacterial irrigant (polymyxinB/bacitracin) and postoperative oral antibiotics (cephalexin, clindamycin, or levofloxacin) in patients undergoing a cardiac implantable electronic devices (CIED) procedure who have at least 2 CIED infection risk factors
Period: Overall Study
Arm/Group | Saline Irrigation | Antibiotic Irrigation and Oral Antibiotics
Started | 505 | 505
Completed | 445 | 445
Not Completed | 60 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Irrigation | Antibiotic Irrigation and Oral Antibiotics | Total
Number analyzed (Participants) | 505 | 505 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.44 (11.2) | 70.42 (11.9) | 70.43 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 146 | 282
  Male | 369 | 359 | 728
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 477 | 470 | 947
  Unknown or Not Reported | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 54 | 107
  White | 433 | 431 | 864
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 17 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 505 | 505 | 1010

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Major Cardiac Implantable Electronic Devices (CIED) Infection
Description: The primary study endpoint will be the number of patients with CIED infection resulting in complete CIED system removal, antibiotic therapy in patients who are not candidates for system removal, or death due to CIED infection.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Irrigation | Antibiotic Irrigation and Oral Antibiotics
Number analyzed (Participants) | 505 | 505
Participants | 5 | 6

2. Secondary Outcome: Number of Patients With a Minor Cardiac Implantable Electronic Devices (CIED) Infection
Description: A minor superficial infection of the incision that does not involve the generator pocket, does not result in any systemic symptoms or signs, and is treated with either observation or a short course of oral antibiotics
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Irrigation | Antibiotic Irrigation and Oral Antibiotics
Number analyzed (Participants) | 505 | 505
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Saline Irrigation | Antibiotic Irrigation and Oral Antibiotics
All-Cause Mortality (participants affected / at risk) | 34/505 | 27/505
Serious Adverse Events (participants affected / at risk) | 5/505 | 6/505
Other Adverse Events (participants affected / at risk) | 245/505 | 218/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Irrigation (N=505) | Antibiotic Irrigation and Oral Antibiotics (N=505)
Infection (Infections and infestations) | 5 (5) | 6 (6) — Infection resulting from surgery or surgical procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Irrigation (N=505) | Antibiotic Irrigation and Oral Antibiotics (N=505)
Tenderness, erythema, or warmth at the pulse generator site (Infections and infestations) | 2 (2) | 1 (1)
Purulent discharge (Infections and infestations) | 4 (4) | 1 (1)
Positive blood culture identifying a coagulase negative staphylococcus (Infections and infestations) | 0 (0) | 1 (1)
Vegetation adherent to CIED hardware (Infections and infestations) | 2 (2) | 2 (2)
Purulent material within pulse generator pocket (Infections and infestations) | 0 (0) | 1 (1)
Allergic Reaction to pouch (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 19 (19) | 20 (20)
Wound hematoma (Surgical and medical procedures) | 22 (22) | 27 (27)
Lead dislodgement (Surgical and medical procedures) | 6 (6) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other device related complication (Product Issues) | 4 (4) | 12 (12)
Other non device related complication (General disorders) | 182 (182) | 149 (149)
Heart transplant (Cardiac disorders) | 2 (2) | 0 (0)
Other (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT02809131/Prot_SAP_000.pdf